CLINICAL TRIAL: NCT03364296
Title: Biological Dating of Cerebral Ischemia With Glutathion S-Transferase-π (GST-π) and Peroxyredoxin 1 (PRDX1) to Detect Patients With Stroke of Unknown Onset Within the Therapeutic Window of Thrombolysis
Brief Title: Biological Dating of Cerebral Ischemia With GST-π/PRDX1 to Detect Patients With Stroke of Unknown Onset Within the Therapeutic Window of Thrombolysis
Acronym: FLAG1
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Dr Sebastien RICHARD, Professor, Central Hospital, Nancy, France
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PHRCI 2016/FLAG1 - RICHARD /MS
Record Dates: First submitted 2017-11-23; First posted 2017-12-06 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Stroke, Acute
Keywords: Acute stroke, Biomarkers
MeSH Terms: conditions — Stroke | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients hospitalized for stroke (Other)
  Interventions: Other: Blood Samples

INTERVENTIONS:
Other: Blood Samples — Blood sample retrieved for biological assessment and biobanking

SUMMARY:
The FLAG1 study will assess the diagnostic performance of biomarkers Glutathion S-Transferase-π (GST-π) and Peroxyredoxin 1 (PRDX1) to identify cerebral infarction of less than 4,5 hours in a population of patients with neurological deficiency of less than 12 hours.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years old
* Patients with symptoms consistent with stroke and a National Institute of Health Stroke Score ≥3 at the inclusion time
* Time symptom onset ≤ 24 hours at inclusion:

  * For patients with time of symptom onset is <4.5h at inclusion, the time of symptom onset has to be precisely known, with a margin of error not exceeding 30 minutes (through patient or witness interview)
  * For patients with time of symptom onset is >4.5h at inclusion, knowledge of precise time of symptom onset is not required. For these patients, to ensure onset-to-inclusion time is between 4.5 and 24 hours at inclusion:
* last time patient presented no deficit must be less than 24 hours,
* symptoms must have been first recognized more than 4.5 hours before blood draw.
* Possibility to perform MRI within the 30 minutes following blood collection
* Person affiliated to or beneficiary of a social security plan

Exclusion Criteria:

* Persons referred in articles L.1121-5, L.1121-7, L.1121-8 and L.1122-2 of the French Public Health Code: Pregnant, parturient or breastfeeding woman ; Minor person (non-emancipated) ; Adult person under legal protection (any form of public guardianship) ; Adult person incapable of giving consent and not under legal protection.
* Persons deprived of liberty for judicial or administrative decision.
* Persons subject to psychiatric care under articles L.3212-1 and L.3213-1 of the French Public Health Code.
* Known cancer in progression.
* Known cirrhosis.
* Myocardial Infarctions, stroke, Subarachnoid hemorrhage or intracranial injury within 3 months prior to enrolment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 930 (Estimated)
Dates: Start 2018-10-15 (Actual); Primary Completion 2024-09-13 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Time (<4.5 hours) between cerebral infarction onset and blood sample for determination for GST-π level | Population will be dichotomized in patients with blood sample performed <4.5 hours and >4.5 hours after stroke onset to determine diagnostic performance of GST-π plasmatic level to identify cerebral infarction of less than 4.5 hours.
  ROC analysis will be performed to determine diagnostic performance (sensitivity, specificity) of GST-π plasmatic level to identify cerebral infarction of less than 4.5 hours.
Time (<4.5 hours) between cerebral infarction onset and blood sample for determination for PRDX1 levels | Population will be dichotomized in patients with blood sample performed <4.5 hours and >4.5 hours after stroke onset to determine diagnostic performance of PRDX1 plasmatic level to identify cerebral infarction of less than 4.5 hours
  ROC analysis will be performed to determine diagnostic performance (sensitivity, specificity) of PRDX1 plasmatic level to identify cerebral infarction of less than 4.5 hours.

SECONDARY OUTCOMES:
Time (<3 and 6 hours) between cerebral infarction onset and blood sample for determination for GST-π and PRDX1 levels | Patient will be dichotomized with blood sample performed <3 and >3 hours, and <6 and >6 hours after stoke onset to determine diagnostic performance of GST-π and PRDX1 plasmatic levels to identify cerebral infarction of less than 3 hours, and < 6 hours
  ROC analysis will be performed to determine diagnostic performance (sensitivity, specificity) of GST-π and PRDX1 plasmatic levels to identify cerebral infarction of less than 3 and 6 hours.
Blood sample for determination for GST-π and PRDX1 levels Cerebral MRI for Diffusion/Perfusion mismatch defining ischemic penumbra | The patient will be included within the 12 hours following stroke onset with one blood sample (defining GST-π and PRDX1 plasmatic levels), and cerebral MRI (defining Diffusion/Perfusion mismatch or penumbra) within the 30 minutes following blood sample.
  ROC analysis will be performed to determine diagnostic performance (sensitivity, specificity) of GST-π and PRDX1 plasmatic levels to identify and quantify ischemic penumbra.
Blood sample for determination for GST-π and PRDX1 levels Cerebral MRI for diagnosis of stroke vs. other diagnosis | The patient will be included within the 12 hours following neurological deficiency onset with one blood sample (defining GST-π and PRDX1 plasmatic levels), and cerebral MRI (defining stroke) within the 30 minutes following blood sample.
  ROC analysis will be performed to determine diagnostic performance (sensitivity, specificity) of GST-π and PRDX1 plasmatic levels to identify stroke.
Blood sample for determination for GST-π and PRDX1 levels Cerebral MRI for diagnosis of ischemic stroke vs. other diagnosis | The patient will be included within the 12 hours following neurological deficiency onset with one blood sample (defining GST-π and PRDX1 plasmatic levels), and cerebral MRI (defining stroke) within the 30 minutes following blood sample.
  ROC analysis will be performed to determine diagnostic performance (sensitivity, specificity) of GST-π and PRDX1 plasmatic levels to identify cerebral infarction.
Blood sample for determination for GST-π and PRDX1 levels Cerebral MRI for diagnosis of hemorrhagic stroke vs. other diagnosis | The patient will be included within the 12 hours following neurological deficiency onset with one blood sample (defining GST-π and PRDX1 plasmatic levels), and cerebral MRI (defining stroke) within the 30 minutes following blood sample.
  ROC analysis will be performed to determine diagnostic performance (sensitivity, specificity) of GST-π and PRDX1 plasmatic levels to identify hemorrhagic stroke.
MRI Diffusion/FLAIR mismatch (yes versus no) | The patient will be included within the 12 hours following stroke onset with one blood sample (defining GST-π and PRDX1 plasmatic levels), and cerebral MRI (defining Diffusion/Perfusion mismatch or penumbra) within the 30 minutes following blood sample.
Volume of cerebral infarction assessed by MRI diffusion weighted imaging. | The patient will be included within the 12 hours following stroke onset with one blood sample (defining GST-π and PRDX1 plasmatic levels), and cerebral MRI (defining Diffusion/Perfusion mismatch or penumbra) within the 30 minutes following blood sample.

CONTACTS AND LOCATIONS:
Locations (5):
- France (5):
  - Centre Hospitalier de Bar-Le-Duc, Bar-le-Duc
  - Hôpital Central, Nancy
  - Fondation Adolphe de Rothschild, Paris
  - Centre Hospitalier de Troyes, Troyes
  - Centre Hospitalier de Verdun, Verdun

REFERENCES:
- [Derived] Karakus A, Girerd N, Sanchez JC, Sabben C, Wietrich A, Lavandier K, Marchal S, Aubertin A, Humbertjean L, Mione G, Bouali S, Duarte K, Reymond S, Gory B, Richard S. Identifying patients with cerebral infarction within the time window compatible with reperfusion therapy, diagnostic performance of glutathione S-transferase-pi (GST-pi) and peroxiredoxin 1 (PRDX1): exploratory prospective multicentre study FLAG-1 protocol. BMJ Open. 2021 Aug 20;11(8):e046167. doi: 10.1136/bmjopen-2020-046167. PMID 34417212